CLINICAL TRIAL: NCT06839300
Title: The International Spinal Cord Injury Blood Biomarker Longitudinal Evaluation (I-SCRIBBLE) Study
Status: Not yet recruiting | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: I-SCRIBBLE
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — 15 mL sample of blood (6 mL for serum, 4 mL for plasma, and 5 mL for RNA isolation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SCI patients: Patients with traumatic SCI
- Non-SCI patients (control group): Non-SCI spine trauma control participants

SUMMARY:
To determine the accuracy of serum NF-L and GFAP levels (ie the biomarkers) at different time points postinjury for predicting the severity of neurologic impairment at 6 months postinjury as either motor complete (AIS grade A/B) or motor incomplete (AIS grade C/D) a group of patients who suffer traumatic spinal fracture and/or dislocation of the spinal column but without neurologic injury will be enrolled as non-SCI spine trauma control participants.

DETAILED DESCRIPTION:
Patients (≥19 years old) with acute blunt non-penetrating traumatic SCI of AIS grade A, B, C, or D will be enrolled at participating sites. The first blood samples will be drawn within 24 hours of injury (the baseline/enrollment visit); afterwards, blood samples are drawn within each successive 24-hour period postinjury until Day 7, and then at 6 months and 12 months postinjury. Blood samples will be drawn from existing lines (eg, arterial line, central venous catheter [CVC] lines, and intravenous [IV] line) that are inserted as part of standard of care. If an existing line has been discontinued, blood will be drawn via venipuncture.

At each time point, one 15 mL sample of blood will be drawn, which will be divided into: 6 mL for serum, 4 mL for plasma, and 5 mL for RNA isolation (for transcriptomics). At any of these time points, an additional 1 mL blood sample will also be drawn for DNA extraction (for the purpose of ApoE genotyping). The samples will first be processed and temporarily stored by the sites and then sent to the coordinating center at UBC, Vancouver, Canada, for central storage and analyses. Levels of NF-L and GFAP in serum and plasma will be analyzed on the Quanterix Simoa instrument (Lexington, KY, US) for each time point collected to determine the accuracy of these biomarkers to stratify injury severity and to predict outcome.

To the extent that is possible, a full ISNCSCI examination will be completed at enrollment. A motor-only exam of the upper and lower extremities will be completed at Day 4 and Day 7 postinjury. A full ISNCSCI examination will be repeated at 6- and 12-month visits. The Spinal Cord Independence Measure (SCIM) version III will be completed at 6- and 12-month visits to assess functional recovery.

A group of patients who suffer traumatic spinal fracture and/or dislocation of the spinal column but without neurologic injury will be enrolled as non-SCI spine trauma control participants. For these participants, one 15 mL sample of blood (6 mL for serum, 4 mL for plasma, and 5 mL for RNA isolation) will be drawn within 24 hours of injury (Day 1) and either at discharge or at Day 7 postinjury, whichever comes first. No additional follow-ups (FUs) are required for these control participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Blunt (non-penetrating) traumatic SCI
* Baseline neurologic impairment deemed "complete" (AIS grade A) or "incomplete" (AIS grade B, C, or D) based on clinical history/examination and/or diagnostic imaging
* Bony spinal level involvement between C0 and L1, inclusive
* Ability to have initial blood sample drawn within 24 hours of injury
* Treated either surgically or non-surgically
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Inclusion criteria for non-spinal cord injury spinal trauma control participants:

* Age ≥ 19 years
* Traumatic spinal fracture and/or dislocation between C0 and L1 (inclusive) without SCI
* Treated either surgically or nonsurgically
* Ability to have initial blood sample drawn within 24 hours of injury
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Penetrating SCI (eg, gunshot, stab)
* Previous SCI
* Isolated spinal injury below L1
* Isolated radiculopathy without fracture
* Isolated cauda equina injury
* Patients with known diagnosis of multiple sclerosis
* Preexisting thromboembolic disease or coagulopathy (disorders related to blood clotting), such as hemophilia or von Willebrand disease
* Patients who in the investigator's opinion will not be compliant with the study procedures and patients who have any other conditions/injuries that in the investigator's opinion would render the study procedures dangerous

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 240 SCI patients with AIS grade A, B, C and D. And 20 non-SCI spine trauma control participants.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of serum NF-L and GFAP biomarkers postinjury for predicting the severity of neurologic imapairement at 6 months postinjury as either motor complete or motor incomplete. | 6 months
  To determine the accuracy of serum NF-L and GFAP levels (ie, the biomarkers) at different time points postinjury for predicting the severity of neurologic impairment at 6 months postinjury as either motor complete (AIS grade A/B) or motor incomplete (AIS grade C/D).
  The primary time points of the serum biomarker levels to be investigated are Day 1, Day 2, Day 3, and Day 4 postinjury (section 5.2). Secondary time points to be explored are Day 5, Day 6, and Day 7 postinjury. These assessment time points also apply to the secondary objectives wherever applicable

SECONDARY OUTCOMES:
Accuracy of serum biomarker levels at different time points postinjury for classifying the baseline injury severity, ie, the AIS grade (A, B, C, and D). | 1 Day - 12 months
  To determine the accuracy of serum biomarker levels at different time points postinjury for classifying the baseline injury severity, ie, the AIS grade (A, B, C, and D).
Accuracy of serum biomarker levels for predicting other neurologic outcomes at 6 months postinjury | 6 months
  To determine the accuracy of serum biomarker levels for predicting other neurologic outcomes at 6 months postinjury. Other neurologic outcomes (apart from the one in the primary objective) include:
  * AIS grade conversion in those with baseline AIS grade A injuries
  * Motor score improvement (ie, ≤ vs > 8-point improvement in total motor score)
Investigate which time point(s) postinjury is/are the most accurate for classifying the baseline AIS grade and predicting neurologic outcomes at 6 months postinjury | 6 months
  To investigate which time point(s) postinjury is/are the most accurate for classifying the baseline AIS grade and predicting neurologic outcomes at 6 months postinjury (ie, motor complete vs motor incomplete, AIS grade conversion, and ≤ vs > 8-point improvement in total motor score).
Investigate whether accuracy of classification and prediction of neurologic outcomes at 6 months postinjury can be enhanced by combining serum NF-L and GFAP levels | 6 months
  To investigate whether accuracy of classification and prediction of neurologic outcomes at 6 months postinjury can be enhanced by combining serum NF-L and GFAP levels.
Investigate whether accuracy of prediction of neurologic outcomes at 6 months postinjury can be enhanced by evaluating the change in serum biomarker levels over time during the first 7 days postinjury. | 6 months
  To investigate whether accuracy of prediction of neurologic outcomes at 6 months postinjury can be enhanced by evaluating the change in serum biomarker levels over time during the first 7 days postinjury.
Investigate the relationship between the accuracy of serum biomarker levels for classification of baseline AIS grade and the perceived reliability of baseline ISNCSCI examination | Baseline
  To investigate the relationship between the accuracy of serum biomarker levels for classification of baseline AIS grade and the perceived reliability of baseline ISNCSCI examination
Determine the accuracy of serum biomarker levels for predicting neurologic outcomes at 12 months postinjury | 12 months
  To determine the accuracy of serum biomarker levels for predicting neurologic outcomes at 12 months postinjury
Determine the accuracy of serum biomarker levels for distinguishing acute traumatic SCI from acute spine trauma without neurologic deficit | Baseline
  To determine the accuracy of serum biomarker levels for distinguishing acute traumatic SCI from acute spine trauma without neurologic deficit via the following:
  * Comparing serum biomarker levels during the first week postinjury between these two groups of patients.
  * Investigating the influence of the severity of spinal column trauma on serum biomarker levels in patients with spine fracture but without neurologic deficit.
Effect of associated trauma on serum biomarker levels | Baseline
  To investigate the effect of associated trauma on serum biomarker levels.
  * Two groups of associated trauma will be investigated: 1) concomitant major injuries to the pelvis, abdomen, chest, or appendicular skeleton, and 2) concomitant TBI.
  * Serum biomarker levels will be compared between patients with and without the two groups of associated trauma.
Relationship between serum and plasma levels of the biomarkers | 12 months
  To investigate the relationship between serum and plasma levels of the biomarkers.
Accuracy of ApoE genotype | 6 and 12 months
  To determine the accuracy of ApoE genotype, ie, presence vs absence of the ApoE ɛ4 allele, for predicting neurologic outcomes at 6 months and 12 months postinjury, either standalone or in combination with the biomarkers
Accuracy of measures of injury severity on baseline MRI | 6 and 12 months
  To investigate the accuracy of measures of injury severity on baseline MRI for classifying baseline AIS grade and predicting neurologic outcomes at 6 months and 12 months postinjury, either standalone or in combination with the biomarkers.
  * To compare the accuracy between MRI measures and serum biomarker levels for classifying baseline AIS grade.
  * To compare the accuracy between MRI measures and serum biomarker levels for predicting neurologic outcomes.
  * To determine whether the accuracy of classification and prediction can be enhanced by combining MRI measures and serum biomarker levels.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kwon, MD, PhD, FRCSC, Principal Investigator — The University of British Columbia

IPD SHARING:
Plan to Share IPD: Undecided